CLINICAL TRIAL: NCT04341168
Title: Clinical and Immunological Characterisation of COVID-19 in Children, Adolescents and Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital of Cologne (Other)
Collaborators: Clinic for Internal Medicine I, University Hospital Cologne, Germany (Unknown); Institute of Virology, University Hospital Cologne, Germany (Unknown); Center for Molecular Medicine Cologne (CMMC) Cologne, Germany (Unknown)
Responsible Party: Principal Investigator, Dr. med. Robert W. Körner, Study Director, University Hospital of Cologne
Other Study IDs: KICC19
Record Dates: First submitted 2020-04-03; First posted 2020-04-10 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — nasopharyngeal swab, oropharyngeal swab, sputum: obtain estimate for viral load of SARS-CoV-2, multiplex PCR for other respiratory viruses, bacterial culture blood: SARS-CoV-2-IgM and -IgG, routine lab values, blood - gas - analysis, blood culture, lymphocyte typing, cytokines, chemokines, HLA-typing, proteome urine: proteome bronchoalveolar lavage: obtain estimate for viral load of SARS-CoV-2, multiplex PCR for other respiratory viruses, bacterial culture, lymphocyte typing, cytokines, chemokines lung biopsy (optional): histology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children and Adolescents with COVID-19: age range: newborn - 18 years old, subgroups will be established
  Interventions: Other: this study is non- interventional
- Adults with COVID-19: age range: from 18 years old, subgroups will be established
  Interventions: Other: this study is non- interventional
- Control group: all ages, any respiratory tract infection, subgroups will be established
  Interventions: Other: this study is non- interventional

INTERVENTIONS:
Other: this study is non- interventional — this study is non- interventional

SUMMARY:
The investigators aim to characterise Coronavirus Disease 2019 (COVID-19) in every age group. On the one hand, emphasis is put on the initial presentation, clinical course, outcome and the therapy used. On the other hand further investigations regarding viral and bacterial coinfections, and response of the immune system will be conducted. This study should serve to improve the understanding of COVID-19, to identify risk factors for a severe clinical course and to obtain further insights into pathophysiology of this new infectious disease.

DETAILED DESCRIPTION:
In 2019 the novel coronavirus severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) was identified as the pathogen causing the Coronavirus Disease 2019 (COVID-19) pandemic. Many retrospective studies have been conducted regarding clinical signs and symptoms and clinical course of the disease. In most cases the infection causes only light symptoms of the upper respiratory tract. The infection can also be asymptomatic. However, in some the disease can cause a severe infection of the lower respiratory tract leading to acute respiratory syndrome (ARDS) which can be fatal. Especially elderly people suffer from severe disease whereas children are less compromised.

In this prospective, monocentric study the investigators include patients of all ages with COVID-19 and also a control group of all ages with respiratory tract infections other than COVID-19. Initial presentation, clinical course, outcome and the therapy used will be recorded. Standard diagnostic procedures (vital signs, results of blood samples, blood gas analysis, x ray, ct scan) will also be recorded. To further characterise the study population naso- and oropharyngeal swabs will be checked for viral and bacterial coinfections. The SARS-CoV-2 viral load will be estimated. To characterise the immunological response IgM- and IgG-antibodies for SARS-CoV-2 will be measured. Moreover lymphocyte typing, cytokine and chemokine analysis will be conducted. The investigators will also include an analysis of the proteome in serum and urine. To characterise the virus-host-interaction HLA analysis of the patients will be conducted. In the case of a medically indicated bronchoscopy bronchoalveolar lavage will be analysed in regards of viral load, coinfections, lymphocyte typing and cytokines / chemokines. In case of a medically indicated lung biopsy or in a post mortem lung biopsy a histological analysis will be made.

In general, samples will be analysed at the initial presentation and after two weeks. Further analysis will be conducted depending on special events like clinical deterioration. Long-term follow up will be ensured by telephone visits.

ELIGIBILITY:
Inclusion Criteria:

* patients with COVID-19: detection of SARS-CoV-2 by PCR in naso- or oropharyngeal swab or sputum, no age limit
* control group: any respiratory tract infection not caused by SARS-CoV-2, no age limit
* informed consent

Exclusion Criteria:

* no respiratory tract infection and no detection of SARS-CoV-2
* no informed consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages either with COVID-19 (symptomatic and asymptomatic) or a respiratory tract infection not caused by SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Clinical course of COVID-19 | 10/2020
  Description of clinical course of COVID-19 in children, adolescents and adults
Analysis of development of antibodies to SARS-CoV-2 | 10/2020
  Measurement of specific IgM- and IgG-antibody production
Estimation of viral load | 10/2020
  Estimation of viral load at initial presentation and after two weeks
Detection of viral coinfections | 10/2020
  A Multiplex PCR will be conducted to test for the most common respiratroy viruses. A naso- and oropharyngeal swab will be used for this
Measurement of cytokine and chemokine response | 12/2020
  Determination of cytokine and chemokine concentrations in serum by ELISA.
Characterisation of virus-host-interaction | 12/2020
  Characterisation of virus-host-interaction by HLA-typing
Identification of disease patterns in proteome | 12/2020
  Identification of disease patterns in proteome by analysis of the proteome in serum and urine
Analysis of change in lymphocyte subtypes | 10/2020
  Detection of change in lymphocyte subtypes in blood and bronchoalveolar lavage
Analysis of histological changes in severe lung disease | 12/2020
  Analysis of histological changes in severe lung disease by lung biopsy
Detection of bacterial coinfections | 10/2020
  A pharyngeal swab will be cultured to check for bacteria residing in the upper airways. Additionally, a blood culture will serve to detect bacteremia

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Körner, Dr., Study Director — Children's University Hospital Cologne; Miguel A Alejandre Alcazar, Prof. Dr. Dr., Study Director — Children's University Hospital Cologne
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No